CLINICAL TRIAL: NCT03612739
Title: An Open-label, Phase I Study to Assess the Safety of NKR-2 Treatment Administered Concurrently With 5-azacytidine in Treatment-naïve Acute Myeloid Leukemia or Myelodysplastic Syndrome Patients Not Candidates for Intensive Therapy
Brief Title: EPITHINK: Epigenetic Drug Treatment and Therapeutic Immunotherapy With NKR-2
Acronym: EPITHINK
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Celyad Oncology SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYAD-N2T-006
Record Dates: First submitted 2018-07-20; First posted 2018-08-02 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2018-11

CONDITIONS: AML, Adult; Myelodysplastic Syndromes
Keywords: CAR-T Cells; NKR-2; AML; Epigenetic drug therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Intervention Model Description: This open-label Phase I study aims to define the recommended dose for further clinical development the NKR-2 treatment administered concurrently with AZA in treatment-naïve AML/MDS patients not candidates for intensive chemotherapy or hematopoietic stem cell transplantation.
  This Phase I study is divided into three sequential cohorts evaluating three different dose-levels of NKR-2 (1x108, 3x108 and 1x109 NKR-2 per injection) using a 3+3 design evaluate. Further patients will be enrolled at the RecD to reach 9 evaluable patients in total at the RecD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 5-azacytidine + 1x10^8 NKR-2 CAR-T Cells
  Interventions: Biological: NKR-2 CAR-T Cells
- Cohort 2 (Experimental): 5-azacytidine + 3x10^8 NKR-2 CAR-T Cells
  Interventions: Biological: NKR-2 CAR-T Cells
- Cohort 3 (Experimental): 5-azacytidine + 1x10^9 NKR-2 CAR-T Cells
  Interventions: Biological: NKR-2 CAR-T Cells

INTERVENTIONS:
Biological: NKR-2 CAR-T Cells — The treatment consists in six consecutive cycles of AZA, administered at days
  1 to 7 of a 28-day cycle. Patients will be treated with 8 injections of NKR-2 at day 9 and 23 of AZA cycles 2-3-4 and 5.
  Other Names: 5-azacytidine (AZA)

SUMMARY:
This open-label Phase I study aims to define the recommended dose for further clinical development the NKR-2 treatment administered concurrently with AZA in treatment-naïve AML/MDS patients not candidates for intensive chemotherapy or hematopoietic stem cell transplantation.

This Phase I study is divided into three sequential cohorts evaluating three different dose-levels of NKR-2 (1x108, 3x108 and 1x109 NKR-2 per injection) using a 3+3 design evaluate. Further patients will be enrolled at the RecD to reach 9 evaluable patients in total at the RecD.

The study consists of a screening phase, a treatment administration phase and a follow-up phase divided into treatment follow-up (TFU) and long-term safety follow-up (LTSFU). For each patient who received at least one NKR-2 administration, the overall study duration will be 15 years after first NKR-2 administration.

DETAILED DESCRIPTION:
This open-label Phase I study aims to define the recommended dose for further clinical development the NKR-2 treatment administered concurrently with AZA in treatment-naïve AML/MDS patients not candidates for intensive induction chemotherapy. The treatment consists in six consecutive cycles of AZA, administered at days

1. to 7 of a 28-day cycle. Patients will be treated with 8 injections of NKR-2 at day 9 and 23 of AZA cycles 2-3-4 and 5.

   This Phase I study is divided into three sequential cohorts evaluating three different dose-levels of NKR-2 (1x108, 3x108 and 1x109 NKR-2 per injection) using a 3+3 design. Further patients will be enrolled at the RecD to reach 9 evaluable patients in total at the RecD. The study consists of a screening phase, a treatment administration phase and a follow-up phase divided into treatment follow-up (TFU) and long-term safety follow-up (LTSFU). For each patient who received at least one NKR-
2. administration, the overall study duration will be 15 years after first NKR-

2 administration. Patients will be asked to complete a total of 54 visits during the treatment administration phase, and 5 visits during the treatment follow-up phase. During the LTSFU, yearly visits will be scheduled (up to Visit Y15).

ELIGIBILITY:
1. The patient must have signed the written ICF and must accept that, beyond the treatment period, and the treatment follow-up period, he/she will have to be monitored for a Long-Term Safety Follow-Up (LTSFU) for up to 15 years after enrollment.
2. Both men and women of all races and ethnic groups are eligible.
3. The patient must be ≥ 18 years old at the time of signing the ICF.
4. The patient must be treatment-naïve with a confirmed diagnosis of either:

4.a. WHO-confirmed de novo or secondary acute myeloid leukemia (AML) with intermediate- or adverse-risk cytogenetics. Note: Patient with AML M3 are excluded. or 4.b. WHO-confirmed myelodysplastic syndrome (MDS) with Revised International Prognostic Scoring System (R-IPSS) criteria [97] for Intermediate, High-risk or Very High-risk (High-grade) disease or refractory anemia with excess blasts (RAEB-1 and RAEB-2).

5. The patient is not eligible for intensive induction chemotherapy. Note: The patient is defined as not eligible for intensive induction chemotherapy on the basis of Investigator's assessment of age, ECOG performance status, comorbidities, regional guidelines, or institutional practice, or all these.

6. The white blood cell-count should be <15x109 cells/L prior to 1st infusion of NKR-2. Note: Use of hydroxyurea (up to C1-D10) is permitted to achieve this concentration (see Section 6.4).

7. The absolute bone marrow blast count should be > 5%. 8. The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2. Note: Patient with anemia resulting in an ECOG performance status 3 is also eligible.

9. The patient must have adequate hepatic and renal functions described in Table 1, as assessed by standard laboratory criteria (with LLN/ULN being the lower/upper limit of normal, respectively): Serum creatinine ≤ 2.0 mg/dL Calculated creatinine clearance > 60 ml/min Total serum bilirubin ≤ 2.0 x ULN Or ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert's Syndrome, hemolysis or transfusion dependence ALT ≤ 3 x ULN AST ≤ 3 x ULN ALT: alanine aminotransferase; AST: aspartate aminotransferase; ULN: upper limit of normal 10. The patient must have a left ventricular ejection fraction (LVEF) of ≥ 40%, as determined by echocardiography or a multigated acquisition (MUGA) scan.

11. The patient must have a good pulmonary function with a Forced Expiratory Volume in the first second (FEV-1)/Forced Vital Capacity (FVC) ≥ 0.7 with FEV-1 ≥ 50% predicted as determined by the spirometry performed at baseline (see Section 7.2.7), unless related to the AML/MDS disease as judged by the Investigator.

12. Women of child-bearing potential and men must agree to use effective contraception before, during and for at least 2 months after the last study treatment administration.

Notes: Adequate contraception is defined as methods of birth control that, alone or in combination, result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. These include established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; male sterilization, true abstinence (when this is in line with the preferred and usual lifestyle of the patient).Women of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as the consequence of hysterectomy, ovariectomy or post-menopause.

13. The patient must, in the opinion of the Investigator, be able to adhere with the study visit schedule and all study procedures described in this protocol.

Exclusion criteria

The patients may not be included in the study if one or more of the following criteria is met:

1. Patients with confirmed or history of tumor involvement in the central nervous system (CNS).
2. Patients who have received any prior AML/MDS therapy (investigational agent or not).

   Note: Patients are authorized to receive hydroxyurea according to specific conditions as detailed in Section 6.4.
3. Patients who are planned to receive, concurrently receiving or have received any investigational agent within 3 weeks before the planned day for the first NKR-2 administration.
4. Patients who are under systemic immunosuppressive drugs, unless specific cases authorized per protocol (see Section 6.4).
5. Presence of any indwelling catheter or drain (e.g., percutaneous nephrostomy tube, indwelling foley catheter, biliary drain, or pleural/peritoneal/pericardial catheter) may be permissible unless they have a catheter-associated infection that cannot be cleared with antibiotics. Ommaya reservoirs and dedicated central venous access catheters such as a Port-a-Cath, peripherally inserted central catheter, or Hickman catheter are permitted.
6. Patients who underwent major surgery within 4 weeks before the planned day for the first NKR-2 administration. Note: Placement of vascular access device is authorized until 10 days before the planned day for the first NKR-2 administration.
7. Patients who have received a live vaccine ≤ 6 weeks prior to each NKR-2 administration.
8. Patients with uncontrolled intercurrent illness or serious uncontrolled medical disorder including, but not limited to evidence of active pneumonitis on screening chest imaging, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia history (or evidenced after the electrocardiogram planned at screening) and/or pronounced disturbances of the electrical conduction system of the heart, or significant thromboembolic events.
9. Patients with significant disorder of coagulation or receiving treatment with warfarin derivatives or heparin.

   Note: Patients receiving systemic individual doses of low molecular weight heparin outside 24 hours prior to each NKR-2 administration are eligible.
10. Patients who have active infections including, but not limited to viral, bacterial or fungal infections necessitating use of antibiotics/antivirals/antifungal treatment (prophylaxis is acceptable).
11. Patients who are known to be positive or screened positive for hepatitis B (HBsAg positive) or C (anti-HCV positive).
12. Patients who are known to be positive or screened positive for the human immunodeficiency virus (HIV).
13. Patients with a family history of congenital or hereditary immunodeficiency.
14. Patients with a history of allergic reactions or hypersensitivity attributed to Human serum albumin, Plasma-lyte A.
15. Patients with a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis and/or active or acute exacerbation of chronic obstructive pulmonary disease (COPD).
16. Patients on supplemental home oxygen.
17. Patients with a history of any autoimmune disease including, but not limited to inflammatory bowel disease (including ulcerative colitis and Crohn's Disease), systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis (e.g.,Wegener's granulomatosis), CNS or motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and myasthenia gravis, multiple sclerosis). Patients with Graves disease and vitiligo will be allowed.
18. Patients with a history of a malignancy other than the one evaluated in this study, with exception of the following circumstances:

    * Patients with a history of malignancy who have been adequately treated and have been disease-free for at least 1 year, and
    * Patients with adequately treated active non-invasive cancers (such as non-melanomatous skin cancer or in-situ bladder, cervical and breast cancers).
19. Patients with psychiatric/social situations or addictive disorders that may compromise the ability of the patients to give informed consent or to comply with the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
The occurrence of Dose Limiting toxicities (DLT) during the study treatment until 6 months after initial treatment. | From Day 1 until the 6 month study visit
  The occurrence of DLTs during the study treatment phase (up to month 6)

SECONDARY OUTCOMES:
Additional Safety Endpoint: the occurrence of Adverse Events and Serious Adverse Events and any toxicity linked to study participation until the end of the administration phase, and until the end of the treatment follow-up. | Study enrollment until the 24 month study visit.
  The occurrence of AEs and SAES and any toxicity linked to study participation until the end of the administration phase, and until the end of the treatment follow up (Month 24).
Overall Survival (OS) Follow-Up | Study enrollment until the 24 month study visit.
  The overall survival (OS), will be evaluated for all patients that received treatment from apheresis until the 24 month study visit.
Relapse-Free Survival (RFS) Follow-Up | Study enrollment until the 24 month study visit.
  The Relapse Free Survival (RFS),patients that do not have an event of Progressive disease, will be evaluated for all patients that received treatment from apheresis until the 24 month study visit.
Event Free Survival (EFS) Follow-Up | Study enrollment until the 24 month study visit.
  The Event Free Survival (EFS), will be evaluated for all patients that received treatment from apheresis until the 24 month study visit.
First Objective Clinical Response | Study enrollment until the 24 month study visit.
  The objective clinical response rate (ORR) post the first NKR-2 administration will be evaluated via bone marrow biopsy and aspirate analysis for disease status.
Duration of First Objective Clinical Response | Study enrollment until the 24 month study visit.
  The duration of response, for patients that achieve complete response or partial response post the first NKR-2 administration will be evaluated for all patients that receive at least the first dose of NKR-2 infusion.
Second Overall Clinical Response | Study enrollment until the 24 month study visit.
  The objective clinical response rate (ORR) post retreatment with NKR-2 administration will be evaluated via bone marrow biopsy and aspirate analysis for disease status.
Duration of Second Overall Clinical Response | Study enrollment until the 24 month study visit.
  The duration of response, for patients that achieve complete response or partial response post the first NKR-2 administration.
Cumulative Incidence of Relapse | Study enrollment until the 24 month study visit.
  The cumulative incidence of relapse (CIR), will be evaluated for all patients that are treated with at least one administration of NKR-2
Cumulative Incidence of Death | Study enrollment until the 24 month study visit.
  The cumulative incidence of Death (CID), will be evaluated for all patients that are treated with at least one administration of NKR-2
Non-relapse Mortality Rate (NMR) | Study enrollment until the 24 month study visit.
  The non-relapse mortality rate (NMR), will be evaluated for all patients that are treated with at least one administration of NKR-2
AML Incidence of Response | Study enrollment until the 24 month study visit.
  For AML patients: the incidence of CR, CRMRD-, CRi, MLFS, PR, or SD post NKR-2 administrations until the end of the treatment follow-up (till 24 months after first NKR-2 treatment administration),
MDS Incidence of Response | Study enrollment until the 24 month study visit.
  For MDS patients: the incidence of CR, PR, marrow CR, cytogenic response, hematologic improvement or SD post NKR-2 administrations until the end of the treatment follow-up (till 24 months after first NKR-2 treatment administration)
Allogeneic Bone Marrow Transplant | Study enrollment until the 24 month study visit.
  The number of patients deemed eligible for an allogeneic stem cell transplantation at screening based on aged and comorbidities by the Investigator who are able to achieve this outcome with investigational treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Lehmann, MD, Study Director — Celyad SA

IPD SHARING:
Plan to Share IPD: Undecided